CLINICAL TRIAL: NCT02634359
Title: Protocol for Evaluation of EarlySense - a Contact-less Heart and Respiration Device for Monitoring Ovulation Cycles and Detection of Early Stages of Pregnancy in Home Environment
Brief Title: Evaluation of EarlySense for Monitoring Ovulation Cycles and Detection of Early Stages of Pregnancy in Home Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ES-CLC-2015_Prot_1_FERT
Record Dates: First submitted 2015-12-14; First posted 2015-12-18 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2018-01

CONDITIONS: Reproduction
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IVF Treatments- Frozen Embryo transfer (Other): Consenting women that arrive to IVF clinic for frozen embryo transfer on spontaneous cycle Study Intervention: Ultrasound and Blood test to detect Ovulation. At home, HR, RR and movements will be contactlessly measured using EarlySense home device
  Interventions: Device: EarlySense home device; Procedure: Vaginal ultrasound; Procedure: Blood Test
- IVF Treatments- Clinical Evaluation (Other): Consenting women that arrive for cycle evaluation or insemination on spontaneous cycle (infertile women).
  Study Intervention: Ultrasound and Blood test to detect Ovulation At home, HR, RR and movements will be contactlessly measured using EarlySense home device
  Interventions: Device: EarlySense home device; Procedure: Vaginal ultrasound; Procedure: Blood Test
- No IVF (Other): Healthy women volunteers with regular menstrual cycles - not using contraceptives Study Intervention: Ultrasound and Blood test to detect Ovulation At home, HR, RR and movements will be contactlessly measured using EarlySense home device
  Interventions: Device: EarlySense home device; Procedure: Vaginal ultrasound; Procedure: Blood Test

INTERVENTIONS:
Device: EarlySense home device — Passive contact-free monitoring at home measuring HR, RR and movements Arms: IVF Treatments- Frozen Embryo transfer IVF Treatments- Clinical Evaluation No IVF
Procedure: Vaginal ultrasound — Vaginal ultrasound for the purpose of determining follicle size Arms:IVF Treatments- Frozen Embryo transfer IVF Treatments- Clinical Evaluation No IVF
Procedure: Blood Test — Hormonal profile blood tests arms: IVF Treatments- Frozen Embryo transfer IVF Treatments- Clinical Evaluation No IVF

SUMMARY:
The study objective is to collect data to assess the accuracy and reliability of Earlysense fertility cycle monitoring performance vs. acceptable known reference methods such as blood tests and intra-vaginal Ultrasound currently used as validated methods to detect ovulation and pregnancy. In addition the collected data will be used to further enhance and improve the existing algorithms.

DETAILED DESCRIPTION:
The study objective is to assess the accuracy and reliability of Earlysense cycle monitoring to detect ovulation and implantation vs. acceptable known reference methods including blood tests and Ultrasound examination that are currently used as validated methods to detect ovulation and pregnancy. In addition the collected data will be used to further enhance and improve the existing algorithms that detect menses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years ≤ 40 years
2. Healthy women with no significant background illness or Consenting women that arrive to IVF clinic for frozen embryo transfer on spontaneous cycle, or Consenting women that arrive for cycle evaluation or insemination on spontaneous cycle (infertile women).
3. Healthy women volunteers with regular menstrual cycles - not using contraceptives
4. Is willing to sign the consent form.
5. Sleeps on a mattress which allows placing a sensor under that mattress(so Earlysense sensor can be inserted under the mattress)
6. Regular cycle

Exclusion Criteria:

* Age < 18 years or > 40 years old
* Is not willing to sign the consent form.
* Does not sleep on a mattress that allows placing EarlySense sensor under it .(e.g., Futon0 Taking any significant medication or have major chronic diseases: e.g. Diabetes, CHF, COPD, Heart disease or pacemaker
* Taking pills (oral contraceptives or medical IUD w. progesterone)
* Women with irregular cycles (PCOS) or un-ovulation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Detecting Ovulation or Early Pregnancy | 3 months
  Determine the effectiveness of the EarlySense system to detect ovulation and early stages of pregnancy. We would like to see what were the differences in measurements on the EarlySense System, on the dates of Ovulation (according to Ultrasound and Blood Test)

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Argaman, Study Director — EarlySense Ltd.
Locations (1):
- Herzelia Medical Center, Herzelia, Israel

IPD SHARING:
Plan to Share IPD: Undecided